CLINICAL TRIAL: NCT01126411
Title: Randomized, Prospective Investigation on the Effects of Immunoadsorption on Pulmonary Vascular Resistance in Patients With Pulmonary Hypertension
Brief Title: Immunoadsorption in Patients With Pulmonary Hypertension
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI left center
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Marcus Doerr, MD, University Medicine Greifswald
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IA-2010-001
Record Dates: First submitted 2010-05-12; First posted 2010-05-19 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Hypertension; Pulmonary Resistance
Keywords: pulmonary hypertension; autoantibodies; immunoadsorption; immunoglobulin substitution; right ventricular function
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): control group / no immunoadsorption
- immunoadsorption (Active Comparator): immunoadsorption
  Interventions: Procedure: immunoadsorption / immunglobulin substitution

INTERVENTIONS:
Procedure: immunoadsorption / immunglobulin substitution — Immunoadsorption with protein-A columns on five consecutive days with subsequent human polyclonal immunoglobulin G substitution after day 5 (0,5g /kg bodyweight)
  Other Names: immunosorba
  Arms: immunoadsorption

SUMMARY:
The purpose of this study is to investigate, if Immunoadsorption of autoantibodies with subsequent substitution of immunoglobulins is able to improve haemodynamics in patients with pulmonary hypertension.

DETAILED DESCRIPTION:
Increased pulmonary precapillary vascular resistance due to vasoconstriction and vasoproliferative processes is the basic pathophysiological mechanism in the development of pulmonary hypertension (PH). In patients with pulmonary arterial hypertension (PH) production of endothelin-1 (ET-1) is increased and elevated ET-1 plasma levels correlate with PH severity As recently shown Autoantibodies against the Endothelin-1 Typ A and Angiotensin II Typ-1 Receptor, which have a high Incidence in PH-Patients, may also play an important role in the pathophysiology of PH (Dandel et al.).

The concept of this study is that the elimination of these autoantibodies by Immunoadsorption with protein A may improve haemodynamics and patient wellbeing. Immunoglobulins are substituted after Immunoadsorption to minimize infection risk.

ELIGIBILITY:
Inclusion Criteria:

* pulmonary hypertension (PH)
* NYHA II-IV
* medical treatment of PH respective to current guidelines
* 18 years or older
* written informed consent of the patient

Exclusion Criteria:

* pulmonary hypertension due to left ventricular dysfunction
* decompensated heart failure
* need for Catecholamines
* active infection
* pregnancy
* malign tumor disease
* other secondary disease with life expectancy < 1 year
* refusal by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
pulmonary vascular Resistance | 3 month
  The extend of change of pulmonary vascular resistance over the observation period will be compared between the 2 groups (treatment versus control group).

SECONDARY OUTCOMES:
echocardiographic parameters: TAPSE | 3 month
  TAPSE=excursion of the lateral tricuspid annulus (measured in m-mode). the extend of cange of TAPSE over the observationperiod will be compared between the 2 groups (treatment vs. controlgroup)
NYHA | 3 month
  NYHA = functional capacity. The extent of change of NYHA-class over the observation period will be compared between the 2 groups (treatment versus control group).
nt pro BNP | 3 month
  nt pro BNP = B-type natriuretic peptide. The extent of change of nt-pro BNP over the observation period will be compared between the 2 groups (treatment versus control group).
peak oxygen uptake (spiroergometry) | 3 month
  The extent of change of peak oxygen uptake over the observation period will be compared between the 2 groups (treatment versus control group).
6 min walktest | 3 month
  The extent of change of 6-min walktest over the observation period will be compared between the 2 groups (treatment versus control group).
ET-1 TYP A Receptor Autoantibody level | 3 month
  The extent of change of ET-1 TYP A Receptor Autoantibody level over the observation period will be compared between the 2 groups (treatment versus control group).
echocardiographic parameters: PAPs | 3 month
  PAPs = systolic pulmonalarterial pressure estimated by maximal flow velocity of tricuspid regurgitant jet (continues doppler).
  The extent of change of PAPs over the observation period will be compared between the 2 groups (treatment versus control group).
electrocardiographic parameters: S´lat. TR Annulus | 3 month
  S´lat. TR Annulus = systolic velocity of the lateral tricuspid annulus measured by tissue doppler.
  The extent of change of S´ lat. TR Annulus over the observation period will be compared between the 2 groups (treatment versus control group).
echocardiographic parameters: AT right ventricular outflow | 3 month
  AT right ventricular outflow = acceleration time of right ventricular outflow, measured by pulsed wave doppler echocardiography.
  The extent of change of AT over the observation period will be compared between the 2 groups (treatment versus control group).

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Ewert, Prof, Study Director — University Medicine Greifswald; Markus Reinthaler, MD, Principal Investigator — University Medicine Greifswald; Lars R Herda, MD, Principal Investigator — University Medicine Greifswald; Stephan B Felix, Prof., Study Chair — University Medicine Greifswald
Locations (1):
- Ernst Moritz Arndt Universität Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany